CLINICAL TRIAL: NCT04614129
Title: Lung Cancer Risk and Early Detection in Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Erica T. Warner, ScD MPH, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020P002693
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer; Lung Diseases
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low-Dose CT (Experimental): Low Dose CT Scan of the Chest
  Interventions: Diagnostic Test: Low Dose CT

INTERVENTIONS:
Diagnostic Test: Low Dose CT — All participants will have a low dose chest CT either within one year of enrollment or after enrollment
  Other Names: LDCT

SUMMARY:
This study will evaluate whether LDCT findings differ between firefighters and non-fighters, the relationship between occupational exposures and LDCT findings, and whether a proteomics assay can further risk-stratify screen-detected nodules among a study population of 850 current and retired firefighters and 1,120 matched controls.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age or with 10 years of firefighting experience
* Current or retired firefighters
* No personal history of lung cancer
* Willing and able to receive LDCT screening at MGH or who have been screened via LDCT within the past year at MGH or another institution, and are willing to release their images to the study

Exclusion Criteria:

* Any active cancer (undergoing treatment or diagnosed within the past 5 years)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Nodule detection rate | 12 months
  Frequency of nodule detection
High-risk nodule detection rate | 12 months
  Frequency of high-risk nodule detection. High risk is defined as a Lung RADS of 3 or 4. Lung RADS categories are as follows: 0) Incomplete; 1) Negative; 2) Benign appearance or behavior; 3) Probably benign; 4) Suspicious

SECONDARY OUTCOMES:
Interstitial lung disease detection rate | 12 months
  Frequency of interstitial lung disease detection
Coronary artery calcification (CAC) ordinal scores | 12 months
  Frequency of high coronary artery calcification (CAC) ordinal scores. Possible scores range from 0 to 12 and high scores are defined as those greater than or equal to 10

CONTACTS AND LOCATIONS:
Overall Officials: Erica T Warner, ScD, Principal Investigator — Massachusetts General Hospital; Lecia V Sequist, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No